CLINICAL TRIAL: NCT05747703
Title: A Telehealth Intervention to Increase Screening and Treatment for Alcohol Use Disorder
Brief Title: Telehealth Treatment for Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ria Health (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Stanford University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1A
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned in a 1:1 to the Ria Treatment Platform or a waitlist control condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ria Treatment Platfrom (Experimental): The Ria Treatment Platform is a telehealth approach that includes medical assessment, prescription of clinically appropriate medications for alcohol use disorder, individual and group coaching, educational video modules, and monitoring of breath alcohol concentrations through a Bluetooth-enabled breathalyzer.
  Interventions: Combination Product: Ria Treatment Platform
- waitlist control (No Intervention): Patients in this arm will not be provided treatment during the study period.

INTERVENTIONS:
Combination Product: Ria Treatment Platform — combined medication, coaching, education, and monitoring
  Arms: Ria Treatment Platfrom

SUMMARY:
Participants with alcohol use disorder will be randomly assigned to either the Ria Treatment Platform or a waitlist control. The Ria Treatment Platform is a telehealth approach that incorporates medical assessment, medications for alcohol use disorder, individual and group coaching, educational video modules, and a Bluetooth-enabled breathalyzer. Patients are followed for three months during which data are collected, including measures of alcohol consumption and its consequences.

ELIGIBILITY:
Inclusion Criteria:

* alcohol use disorder

Exclusion Criteria:

* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
percent of subjects without heavy drinking | last four weeks
  percent of subjects without heavy drinking per timeline follow-back

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — Ria Health
Locations (1):
- Stanford University, Stanford, California, United States